CLINICAL TRIAL: NCT02364128
Title: Patient-Centered Outcomes Research Institute (PCORI)- Improving Patient Decisions About Bariatric Surgery
Brief Title: Improving Patient Decisions About Bariatric Surgery
Acronym: PCORI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Amir Ghaferi, Assistant Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00083670
Record Dates: First submitted 2015-01-22; First posted 2015-02-16 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Morbid Obesity; Weight Reduction
MeSH Terms: conditions — Obesity, Morbid; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Potential bariatric surgery patients who receive both the baseline questionnaire and follow-up questionnaire.
- Decision Aid (Other): Potential bariatric surgery patients who receive both the baseline questionnaire decision aid/conjoint analysis and follow-up questionnaire.
  Interventions: Behavioral: Decider Guider: Weight Loss

INTERVENTIONS:
Behavioral: Decider Guider: Weight Loss — Decision aid tool about weight loss treatment
  Arms: Decision Aid

SUMMARY:
At least 15 million Americans are morbidly obese, or more than 100 pounds overweight. Medical treatments including drugs and behavior modification have proven ineffective in producing significant and lasting weight loss in this group. While bariatric surgery is extremely effective for most patients, it also carries risks for both short and long-term complications. There are currently four different types of bariatric surgery available and the risks and benefits of these procedures vary widely and are strongly affected by patient and clinical characteristics.

Decision making under these circumstances should reflect informed patient's values and preferences regarding these trade-offs. Instead, the choice of bariatric procedure is more often driven by the beliefs and experiences of the bariatric surgeon that a patient happens to see. Variability in the type of surgery recommended to patients likely results from some combination of surgeons' subjective opinions and personal experiences with regard to the risks and benefits of the treatment options and delegated decision making on the part of patients.

The goals of this research proposal are to develop, implement, and evaluate an informed decision support tool for treatment of morbid obesity. This project will be conducted within the context of the Michigan Bariatric Surgery Collaborative (MBSC), which is a statewide clinical registry and quality improvement program that has the participation of virtually every bariatric surgeon and program in the state of Michigan. The MBSC registry now includes externally audited clinical data for more than 80,000 consecutive bariatric surgery patients. MBSC outcome measures include complications occurring within 30 days as well as weight loss, comorbidity resolution, quality of life and satisfaction at 1, 2, and 3 years after bariatric surgery.

DETAILED DESCRIPTION:
Our specific aims are:

1. To develop a web-based interactive decision support tool to incorporate tailored information regarding risks and benefits of the treatment options (from regression-based prediction models derived on the 35,000 patients already in the MBSC registry) with information regarding other salient attributes of the treatment options (derived from focus groups and semi-structured interviews with stakeholders including bariatric surgery patients, bariatric program staff, and surgeons).
2. To perform a quasi-experimental study comparing the decision support tool with usual care to determine its effects on patient decisions (treatment choice, knowledge, treatment-preference concordance, and decisional conflict) and on patient outcomes including weight loss, patient satisfaction, and improvements in quality of life after surgery.

This research is closely aligned with the goals of PCORI and will have direct impacts on patients and caregivers by providing information that is required to improve healthcare decision-making for this prevalent, damaging, and costly condition.

ELIGIBILITY:
Inclusion Criteria:

* All patients considering undergoing bariatric surgery in the state of Michigan who are 18 or older.
* All patients, regardless of gender or racial/ethnic background, will be recruited to participate in the study in the same way.

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
Decision outcome by Decider Guider Questionnaire | 24 months
  Decisional measures
Patient specific outcome by Decider Guider Questionnaire | 24 months

SECONDARY OUTCOMES:
Knowledge, as measured by a follow-up Decider Guider questionnaire to test knowledge | 24 months
Preferences as measured by Decider Guider Questionnaire | 24 months
Weight | 24 months
Quality of Life as measured by Decider Guider Questionnaire | 24 months
Comorbidity Resolution as measured by Decider Guider Questionnaire | 24 months
Patient Satisfaction as measured by Decider Guider Questionnaire | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States